CLINICAL TRIAL: NCT05336773
Title: Research on Artificial Intelligence-based Mayo Score Recognition System for Disease Activity Degree of Ulcerative Colitis Under Digestive Endoscopy
Brief Title: Ulcerative Colitis Mayo Score With Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yanling Wei, Associate chief physician, M D., Third Military Medical University
Other Study IDs: TMMU-DP--002
Record Dates: First submitted 2022-02-27; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis; Colonoscopy; Deep Learning
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will use deep learning to classify colonoscopy images of different severity of ulcerative colitis, so as to assist clinicians in the accurate diagnosis of ulcerative colitis.

DETAILED DESCRIPTION:
In this project, artificial intelligence was used to colonoscopic images of patients with ulcerative colitis with different disease activity levels and classify them according to the evaluation standard Mayo score to assist endoscopists in identifying disease activity levels of patients with ulcerative colitis during colonoscopy. It can help clinical endoscopists to accurately identify, and the visualization technology of artificial intelligence category response map can comprehensively display the areas with high importance for deep network classification results, and visualize the experimental lesion sites, thus effectively verifying the reliability and interpretability of deep network. This study can provide strong support for accurate identification of disease activity in clinical ulcerative colitis, effectively reduce the workload of clinicians, and provide a convenient, effective and practical clinical teaching tool.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were 18-72 years old, male and female;
2. Clinical diagnosis of ulcerative colitis;
3. The subjects underwent colonoscopy and the colonoscopy report was complete.

Exclusion Criteria:

1. Subjects are younger than 18 years old or older than 72 years old;
2. Subjects underwent colectomy, ileostomy, colostomy, ileostomy, or other intestinal resection;
3. subjects with ambiguous diagnosis.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The images were retrieved from the endoscopy database of Army Medical Center of PLA and obtained from the colonoscopy of patients with ulcerative colitis who met the inclusion criteria. The data images were used to establish and verify the model of ai-assisted recognition system.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The accuracy of deep learning model in the training and validation datasets assessment of Mayo score in ulcerative colitis patients. | Through study completion, an average of 1 year.
  In the training and validation datasets, we plotted the AUC (area under curve) for Mayo 0, Mayo 1, Mayo 2, and Mayo 3 to evaluate our model objectively.

SECONDARY OUTCOMES:
The accuracy and time efficiency of endoscopists assessment of Mayo score in ulcerative colitis patients. | Through study completion, an average of 1 year.
  The dataets were randomly assigned to endoscopists. All endoscopists were trained in diagnostic studies, finished both clinical and specific endoscopic training, and were not involved in the enrollment and labeling of the patients and images. During the comparison test, all data were randomized and deidentified beforehand. The average time spent by 10 endoscopists in diagnosing the test dataset in the deep learning model and the number of correct cases were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yanling Wei, Professor, Study Director — Third Military Medical University
Locations (1):
- Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Qi J, Ruan G, Ping Y, Xiao Z, Liu K, Cheng Y, Liu R, Zhang B, Zhi M, Chen J, Xiao F, Zhao T, Li J, Zhang Z, Zou Y, Cao Q, Nian Y, Wei Y. Development and validation of a deep learning-based approach to predict the Mayo endoscopic score of ulcerative colitis. Therap Adv Gastroenterol. 2023 May 22;16:17562848231170945. doi: 10.1177/17562848231170945. eCollection 2023. PMID 37251086